CLINICAL TRIAL: NCT06840509
Title: BIO|CONCEPT.CorSky Family, First in Human Study for the CorSky ICD Family
Brief Title: BIO|CONCEPT.CorSky, First in Human Study for the CorSky ICD Family
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik Australia Pty Ltd. (Industry)
Collaborators: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Organization: Biotronik SE & Co. KG (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TA120
Record Dates: First submitted 2025-02-18; First posted 2025-02-21 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-02

CONDITIONS: Tachycardia; Heart Failure
MeSH Terms: conditions — Tachycardia; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with indication for ICD or CRT-D therapy according to standard clinical guidelines. (Experimental)
  Interventions: Device: CorSky ICD or CRT-D

INTERVENTIONS:
Device: CorSky ICD or CRT-D — Subjects with an indication for an ICD or CRT-D device will be implanted with a CorSky device of the CorSky ICD family according to standard implantation procedures. Device programming will be done according to the medical needs of the subjects.

SUMMARY:
The goal of this exploratory study is to test the preliminary safety and product performance of the new CorSky ICD family in subjects that require an ICD or cardiac resynchronization therapy with defibrillation (CRT-D). The study will be conducted at sites in Australia and New Zealand. It is planned to include 50 subjects in the study. Participants will visit sites at enrollment in the study, at implantation, pre-hospital discharge, 1- 3- and 12-month follow-up visits. At the visits the device will be interrogated and standard device measurements including those related to special features will be performed to assess the functionality of the device. Programming of the ICDs will be done according to the participant´s therapeutical needs.

ELIGIBILITY:
Inclusion Criteria:

* Standard indication for ICD or CRT-D therapy according to clinical guidelines
* Planned for de novo implantation of an ICD/CRT-D, or upgrade/exchange from existing ICD/CRT-D or pacemaker implant
* Ability to understand the nature of the study
* Willingness to provide written informed consent
* Ability and willingness to perform all on-site follow-up visits at the study site Ability and willingness to use the CardioMessenger and acceptance of the BIOTRONIK Home Monitoring concept

Exclusion Criteria:

* For VR-T DX and CRT-DX: Permanent atrial tachyarrhythmia
* For VR-T DX and CRT-DX: Patients requiring atrial pacing
* Planned for His-Bundle-Pacing
* Planned cardiac surgical procedures or interventional measures other than the study procedure within the next 12 months
* Pregnant or breast feeding
* Age less than 18 years
* Participation in another interventional clinical investigation according to the definition given below 2,3
* Life-expectancy less than 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Serious adverse device effect (SADE)-free rate after 12 months | 12 months
  Descriptive statistics of the investigational device related SADE-free rate after first implantation attempt will be calculated using a Kaplan-Meier estimate

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Alexandra Hospital, Brisbane, Australia

IPD SHARING:
Plan to Share IPD: Undecided